CLINICAL TRIAL: NCT02611284
Title: Less Invasive Beractant Administration in Preterm Infants: a Pilot Study.
Brief Title: Less Invasive Beractant Administration in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Manuel Sanchez Luna, Dr, Hospital General Universitario Gregorio Marañon
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-01
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Infant, Premature
Keywords: Beractant; Feasibility Studies; Infant, Premature; Noninvasive Ventilation
MeSH Terms: conditions — Premature Birth | interventions — Insure Cement

ARMS (2):
- Treatment Cohort (LISA) (Experimental): All preterm infants born at < 32 WG between October 2013 and November 2014 who met inclusion criteria were managed by the new LISA technique.
  Interventions: Procedure: LISA
- Historical Cohort (INSURE) (Other): The control group was collected from the period immediately before the study's initiation (from Jun 2012 to September 2013). This cohort was comprised of preterm infants of less than 32 WG who met the inclusion criteria.
  Interventions: Procedure: INSURE

INTERVENTIONS:
Procedure: LISA — All infants were supported with nCPAP while breathing spontaneously during instillation. A 5Frenchgamma sterilized multi-access catheter specifically designed to deliver surfactants for Neonates was placed 1-2 cm below the vocal cords by direct laryngoscopy without the use of a Magill forceps. Beractant was used as exogenous natural surfactant, (100mg/kg; 4ml/kg) and administered in two aliquots during 1-3 minutes. Positive pressure inflations were given by a mask and bag only if the infant was apneic or bradycardia develops despite the interruption of the procedure. The surfactant administration catheter was removed after surfactant instillation and nCPAP support was maintained. A second dose of surfactant was administered during the first 3 days of life if more than 40% of FiO2 was needed while on nCPAP with at least 6 cm H2O pressure.
  Arms: Treatment Cohort (LISA)
Procedure: INSURE — The INSURE technique was performed using Beractant (4ml/kg) after endotracheal intubation. A multi-access catheter for Neonates/Pediatrics designed to deliver surfactants (KimVentTrach Care Technology ®, United Kingdom) was pre-connected to the endotracheal tube and used for surfactant administration without having to disconnect the ventilator. While surfactant was administered all infants were connected to pressure support ventilation modality (PSV) combined with volume guarantee (VG), Dräger ventilator). A tidal volume of 4ml/kg was initially adjusted.
  After surfactant administration, all infants were to be extubated, in accordance with our institutional extubation guidelines, if FiO2< 0.35; for a target Oxygen Saturation (SpO2) of >90%, and if a consistent respiratory effort was present. Extubation was supported with nCPAP in all patients.
  Arms: Historical Cohort (INSURE)

SUMMARY:
The aim of this study is to assess the efficacy and feasibility of a new less invasive surfactant administration (LISA) technique with a specific designed cannula for surfactant administration using Beractant replacement in preterm infants <32 weeks of gestation and compare short and long term outcomes with the intubation, administration of surfactant and extubation method (INSURE).

This was a single-center, prospective, open-label, non-randomized, controlled study with an experimental cohort of 30 patients treated with LISA and a retrospective control group comprising the 30 most recently treated patients with INSURE. Beractant (4 ml/Kg) was administered as exogenous surfactant in both groups if patients on nasal continuous positive airway pressure (nCPAP) during the first three days of life were needed of more than 30% of fraction of inspired oxygen inspired oxygen fraction (FiO2).

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants of less than 32 weeks of gestation (WG)breathing spontaneously on nCPAP during the first three days of life that met exogenous surfactant administration criteria (Table l) were eligible to enroll in the study

Exclusion Criteria:

* Infants who met intubation criteria (Table 1) at the moment of the surfactant administration were excluded in both groups.

Ages: 1 Minute to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
% patients >1 h of mechanical ventilation | through study completion, an average of 1 year
  The percentage of patients that required more than 1 hour of mechanical ventilation during the first three days of age.

SECONDARY OUTCOMES:
need for intermittent mechanical ventilation (iMV) | through study completion, an average of 1 year
  need for iMV at any time and its duration
second dose of surfactant | through study completion, an average of 1 year
  the requirement of a second dose of surfactant
bradycardia episodes | through study completion, an average of 1 year
  the number of bradycardia episodes (<100 bpm) needing pressure inflations (PPI) during instillation
attempts to catheterize | through study completion, an average of 1 year
  the number of attempts to catheterize the trachea was recorded
surfactant reflux cases | through study completion, an average of 1 year
  the number of surfactant reflux cases

REFERENCES:
- [Derived] Ramos-Navarro C, Sanchez-Luna M, Zeballos-Sarrato S, Gonzalez-Pacheco N. Less invasive beractant administration in preterm infants: a pilot study. Clinics (Sao Paulo). 2016 Mar;71(3):128-34. doi: 10.6061/clinics/2016(03)02. PMID 27074172